CLINICAL TRIAL: NCT04551339
Title: Zinc Versus Multivitamin Micronutrient Supplementation to Support Immune Health in the Setting of COVID-19 Pandemic: A Randomized Study
Brief Title: Zinc Versus Multivitamin Micronutrient Supplementation in the Setting of COVID-19
Acronym: ZnCOVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Atta Behfar, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-004637
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Healthy; Health Care Worker Patient Transmission; Aging
Keywords: Zinc; Immune health
MeSH Terms: interventions — Tablets; Geritol; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose Zinc (PreserVision AREDS formulation soft gels or tablets) (Active Comparator): Subjects will have a high dose Zinc supplementation in combination with Copper, Vitamin C/E and beta-carotene
  Interventions: Dietary Supplement: PreserVision AREDS formulation soft gels or tablets
- Multivitamin with 11mg of zinc (Active Comparator): Subjects in this arm will have a multivitamin supplement with 11mg of zinc
  Interventions: Dietary Supplement: Multivitamin with 11mg of zinc

INTERVENTIONS:
Dietary Supplement: PreserVision AREDS formulation soft gels or tablets — Two tabs taken daily for three months
  Arms: High dose Zinc (PreserVision AREDS formulation soft gels or tablets)
Dietary Supplement: Multivitamin with 11mg of zinc — One tab taken daily for three months
  Arms: Multivitamin with 11mg of zinc

SUMMARY:
The purpose of this research study is to look at high dose zinc versus multivitamin micronutrient supplementation to support immune health in the setting of the COVID-19 pandemic.

DETAILED DESCRIPTION:
This is a two-cohort prospective randomized study intended to test the role of Zinc versus multivitamin supplementation in supporting immune health in the setting of the COVID-19 pandemic. Individuals over 50 years old or primary health care professionals over the age of 18 who have had no evidence of prior COVID-19 infection and who have been asymptomatic for 7 days prior to enrollment will be randomized at the individual level to take either PreserVision AREDS formulation soft gels or tablets with 69.6mg/day Zinc supplementation or to receive a multivitamin supplement with 11mg of zinc/day.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years old OR primary healthcare professional (defined as having a job that has had direct patient contact during the COVID-19 pandemic) and ≥18 years old
* No symptoms of COVID-19 (a fever of 100.0o F or greater, OR a new cough, OR new shortness of breath, OR new sore throat, OR new diarrhea, OR new fast breathing (respiratory distress), OR new chills, OR new muscle aches (myalgias), OR new loss of smell, OR new change or loss of taste sensation) in the past 7 days
* Have a negative Elecsys Anti-SARS-CoV-2 immunoassay antibody test at screening
* Have not had close contact with a person with a LABORATORY CONFIRMED case of COVID-19 without full PPE (Close contact is defined by CDC as: Being within approximately 6 feet of a COVID-19 patient for a total of 15 minutes or more over a 24 hour period) or having direct contact with infectious secretions of a COVID-19 patient (e.g. being coughed on)) in the last 14 days
* Mayo Clinic patient who has a patient online account set up or is willing to set up an online account
* Must have a valid email address and internet service

Exclusion Criteria:

* History of positive or indeterminate COVID PCR test prior to screening or Elecsys Anti-SARS-CoV-2 immunoassay antibody test positive or indeterminate at screening
* Active symptoms of COVID ((a fever of 100.0o F or greater, OR a new cough, OR new shortness of breath, OR new sore throat, OR new diarrhea, OR new fast breathing (respiratory distress), OR new chills, OR new muscle aches (myalgias), OR new loss of smell, OR new change or loss of taste sensation)) in past 7 days
* Known intolerance to multivitamins or zinc supplements from prior exposure
* Inability to complete follow-up questions or grant access to electronic health record for surveillance
* Have had close contact with a person with a LABORATORY CONFIRMED case of COVID-19 in past 14 days
* Current or former smoker less than 5 years ago
* Pregnant or breastfeeding
* Prisoner
* Any subject with known immunosuppressed state, including

  1. A history of solid organ or bone marrow transplantation
  2. Subjects currently receiving chemotherapy
  3. Current rheumatologic or autoimmune illness requiring treatment with glucocorticoids, antimetabolite agents (methotrexate, azathioprine, mercaptopurine, fluorouracil, mycophenolate, leflunomide), IMIDs (lenalidomide, thalidomide, pomalidomide), calcineurin inhibitors (tacrolimus, cyclosporine), mTOR inhibitors (sirolimus, everolimus), or any monoclonal antibody drugs (including any drug given intravenously or subcutaneously) for the purpose of immunosuppression
  4. Subjects with HIV or primary immunodeficiency syndromes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
COVID-19 illness requiring hospitalization | Through study completion, approximately 3 months
  Total number of subjects admitted to the hospital in relations to COVID-19 illness PCR or undergo seroconversion

SECONDARY OUTCOMES:
Illness without hospitalization | Through study completion, approximately 3 months
  Total number of subjects with COVID-19 illness that are not hospitalized
Supplemental oxygen therapy during hospitalization | Through study completion, approximately 3 months
  Total number of subjects to require supplemental oxygen therapy during hospitalization for COVID-19
Invasive ventilation during hospitalization | Through study completion, approximately 3 months
  Total number of subjects to require invasive ventilation during hospitalization for COVID-19
Mortality | Through study completion, approximately 3 months
  Total number of subject deaths

CONTACTS AND LOCATIONS:
Overall Officials: Atta Behfar, MD, PhD, Principal Investigator — Mayo Clinic; Albert Hakaim, MD, Principal Investigator — Mayo Clinic; Ayan Sen, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Scottsdale, Scottsdale, Arizona
  - Mayo Clinic in Jacksonville, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota